CLINICAL TRIAL: NCT00837174
Title: Phase II Study of Combination Vorinostat and Bortezomib in Patients With Relapsed and/or Refractory Non-Hodgkin Lymphoma
Brief Title: Relapsed and/or Refractory Non-Hodgkin Lymphoma Study
Acronym: COMBOSTAT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never activated/opened as funding source and other support not available.
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00002085; 0908-0284 (Other: Houston Methodist Research Institute IRB)
Record Dates: First submitted 2009-02-03; First posted 2009-02-05 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: non-Hodgkin Lymphoma; aggressive lymphoma; indolent lymphoma; B cell lymphoma; T cell lymphoma; Diffuse large B cell lymphoma; anaplastic large B cell lymphoma; lymphoblastic lymphoma; Burkitt's lymphoma; transformed follicular center cell lymphoma; transformed marginal zone lymphoma; transformed small lymphocytic lymphoma; grade 3 follicular center cell lymphoma; blastic form marginal zone lymphoma; transformed cutaneous T cell lymphoma; mycosis fungoides stage IV; angioimmunoblastic lymphadenopathy-like T-cell lymphoma; nasal NK/T cell lymphoma; peripheral T-cell lymphoma; small lymphocytic lymphoma; lymphoplasmacytic lymphoma; follicular center cell lymphoma grade 1; follicular center cell lymphoma grade 2; mantle cell lymphoma; marginal zone lymphoma; mycosis fungoides
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, T-Cell; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Mycosis Fungoides; Lymphoma, T-Cell, Peripheral; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell | interventions — Vorinostat; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Vorinostat + Bortezomib (Experimental): Six cycle combination therapy with vorinostat and bortezomib.
  Interventions: Drug: Vorinostat in combination with Bortezomib

INTERVENTIONS:
Drug: Vorinostat in combination with Bortezomib — Patients will be treated with oral vorinostat on days 1 through 14 followed by a 7-day rest period, for a 21-day treatment cycle for up to 6 cycles in the absence of disease progression or unacceptable toxicity. The patients will receive once-daily oral vorinostat (400 mg) with bortezomib 1.3 mg/m2 as an IV push on days 1, 4, 8, 11.
  Other Names: vorinostat (Zolinza); bortezomib (Velcade)

SUMMARY:
The purpose of this study is to determine the rate of response to the drugs bortezomib (Velcade) and vorinostat (Zolinza), when used in combination, in patients with relapsed (recurrent) and/or refractory (difficult to treat) non-Hodgkin Lymphoma, and to determine the safety and tolerability of this regimen.

DETAILED DESCRIPTION:
More selective and less toxic therapeutic strategies are needed to improve cure rates and prolong survival in patients with relapsed and/or refractory non-Hodgkin Lymphoma.

Amongst the multiple new pathways recently studied two have emerged as potentially important targets for new agents in lymphoma. These include the ubiquitin proteasome pathway and the biochemical reactions that control histone acetylation. The first two agents in each class to have been studied in lymphomas are: bortezomib and vorinostat. Bortezomib has been granted FDA approval for the treatment of mantle cell lymphoma and has established activity in a variety of B-cell lymphomas including follicular, marginal zone and diffuse large B-cell lymphoma. Vorinostat or SAHA (suberoylanilide hydroxamic acid) has been FDA approved for the treatment of refractory cutaneous T-cell lymphomas and has also shown activity in other lymphomas.

Synergistic activity between vorinostat and bortezomib has been observed in different cell lines. The proposed study will be a phase II trial of the combination of vorinostat and bortezomib at the recommended dose-schedule in patients with recurrent and/or refractory lymphomas, indolent and aggressive, and B or T.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-Hodgkin Lymphoma including small lymphocytic lymphoma, lymphoplasmacytic lymphoma, follicular center cell lymphoma, mantle cell lymphoma, marginal zone lymphoma, diffuse large B cell lymphoma, Burkitt's lymphoma, lymphoblastic lymphoma, anaplastic large cell lymphoma, nasal NK/T cell lymphoma, mycosis fungoides/Sezary syndrome, angioimmunoblastic T-cell lymphoma and peripheral T-cell lymphomas not otherwise specified
* Received 2 or > prior therapies, which may include hematopoietic cell transplant (HCT)
* Received treatment with a nucleoside analog, or an alkylating agent, an anthracycline and/or in the case of B cell lymphomas, rituximab
* Resistant disease to 2 regimens or resistant disease to at least 1 regimen after first relapse
* Bi-dimensionally measurable disease documented within 30 days prior to enrollment. Bidimensionally measurable disease is defined as:

  * A lymph node or tumor mass that can be accurately measured in two dimensions by CT,MRI, medical photograph (skin or oral lesion), plain X-ray, PET scan or other conventional technique and a greatest diameter of 1 cm or >; or palpable lesions with both diameters > 2 cm (lesion measured in 2 largest perpendicular dimensions in millimeters)
  * For the purposes of this protocol, disease should be located in an area of no prior radiation therapy or a clear progression in an area that was previously irradiated
* Adequate organ and marrow function obtained < or = to 14 days prior to enrollment as defined by a(n):

  * ANC > or = to 1,000/microliter
  * Platelet count > or = to 100,000/microliter, or > or = to 75,000/microliter if the bone marrow is involved
  * Hemoglobin level > or = to 9 g/dL
  * Total bilirubin < or = to 1.5 x institutional upper limit of normality (ULN).(If abnormal, direct bilirubin less than or equal to 1.5 x institutional ULN)
  * ALT or AST < or = to 2.5 x institutional ULN (< or = to 5 x institutional ULN if liver involvement with lymphoma)
  * Serum creatinine < or = to 1.5 x institutional ULN
* Zubrod (ECOG) Performance Status of 0 or 1
* Age > than or = to 18 years
* Life expectancy > or = to 3 months as clinically determined by referring physician
* Female patient is either post menopausal, free from menses for > 2 years, surgically sterilized or willing to use highly effective methods of contraception (i.e., a condom in conjunction with a diaphragm, or spermicidal jelly; or oral, injectable, or implanted birth control; or abstinence ) to prevent pregnancy throughout the study, starting with visit 1
* Female patients of childbearing potential must have a negative serum pregnancy test (beta-HCG) within 72 hours of enrollment and should not be nursing due to the potential for congenital abnormalities and of harm to nursing infants due to this treatment regimen
* Male patient agrees to use an adequate method of contraception (i.e., a condom if female partner uses a diaphragm, spermicidal jelly; or oral, injectable, or implanted birth control; or abstinence) for the duration of the study and for 12 weeks after the last dose
* Patient must be able to swallow capsules
* Signed and dated IRB/ethics committee-approved informed consent before any protocol specific screening procedures are performed
* Both men and women of all races and ethnic groups are eligible for this trial

Exclusion Criteria:

* Prior investigational therapy within 3 weeks of enrollment. Investigational therapy is defined as treatment that is not approved for any indication
* CNS metastases, as indicated by clinical symptoms,cerebral edema, requirement for corticosteroids and/or progressive growth (treated CNS metastases must be stable for greater than 2 weeks prior to enrollment)
* Active second malignancy that requires treatment or that would interfere with assessment of response
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer with < 5 years of documented disease-free status
* Treatment with the following within the timeframe specified prior to enrollment:

  * Chemotherapy, radiotherapy, immunotherapy (active (such as vaccines) or passive (such as monoclonal antibodies or immunotoxins)) or major surgery < or = to 3 weeks;
  * Nitrosourea, or mitomycin < or = to 6 weeks
  * Radioimmunotherapy (e.g. Bexxar or Zevalin) < or = to 12 weeks
  * Concurrent enzyme-inducing anticonvulsant agents or valproic acid in last 4 weeks
  * Prior bortezomib or any other proteasome inhibitor
  * Prior vorinostat or any other histone deacetylase inhibitor
  * Concurrent systemic corticosteroids (<10 mg/day of prednisone or equivalent for adrenal insufficiency or acute allergic reactions allowed)
* Uncontrolled current illness including, but not limited to:

  * Clinically or laboratory determined active infection
  * Clinically limiting congestive heart failure or ejection fraction (EF) <45%
  * Clinically unstable angina pectoris (or myocardial infarction within 6 months of Day 1)
  * Clinically significant cardiac arrhythmia
  * Limiting pulmonary hypertension
  * Pre-existing neuropathy ≥ grade 2
  * Patients with pleural effusions, ascites or peripheral edema grade 2 or >
* HIV
* Active viral hepatitis
* Major surgery or significant traumatic injury within 21 days prior to enrollment (this does not apply to placement of a venous access device)
* Hypersensitivity to any of the components in vorinostat or bortezomib or agents containing boron or mannitol
* Significant psychiatric illness/social situations that would limit compliance with study medication and requirements of the study as determined by study MD
* Significant medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the subject's risk by participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Determine the response rate of this regimen in this patient population. | 6 cycles

SECONDARY OUTCOMES:
Determine the progression free survival of this regimen in this patient population. | entire length of study
Determine the safety and tolerability of this regimen in this patient population. | throughout course of study
To correlate response rate and progression free survival with pre-treatment and post-treatment NFkB, TRAIL, cyclin D1, histone acetylation, EBV related proteins, and CTA expression. | 6 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Hector A Preti, M.D., Principal Investigator — The Methodist Hospital Research Institute

IPD SHARING:
Plan to Share IPD: Undecided
To be determined